CLINICAL TRIAL: NCT01479101
Title: Prospective Neo-adjuvant REGISTRY Trial Linking MammaPrint, Subtyping and Treatment Response: Neoadjuvant Breast Registry - Symphony Trial (NBRST) (Pronounced "in Breast")
Brief Title: NBRST: Prospective Neo-adjuvant REGISTRY Trial
Acronym: NBRST
Status: Completed | Type: Observational
Sponsor: Agendia (Industry)
Responsible Party: Sponsor
Other Study IDs: P0339 NBRST Registry
Record Dates: First submitted 2011-11-18; First posted 2011-11-24 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer
Keywords: neo adjuvant, breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — As part of routine breast cancer treatment, the doctor will conduct a core needle biopsy and provide tissue from the tumor to Agendia for testing. After the diagnostic test(s) from the Agendia Breast Cancer Suite have been performed on the tumor specimen, there might be some remaining tissue left.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MammaPrint, BluePrint, neo-adj CT or HT: All patients receive the MammaPrint and BluePrint gene expression profile. Treatment at the discretion of the physician while adhering to NCCN guidelines.
  Interventions: Other: MammaPrint 70-gene expression profile; Other: BluePrint 80 gene expression profile

INTERVENTIONS:
Other: MammaPrint 70-gene expression profile
Other: BluePrint 80 gene expression profile

SUMMARY:
The scope of this registry study is to measure chemosensitivity as defined by pCR (primary endpoint), or endocrine sensitivity as defined by partial response (decrease in longest tumor diameter or residual cancer burden category 1 (RCB1), a primary endpoint for neo-adjuvant endocrine therapy and a secondary endpoint for neoadjuvant chemotherapy), metastasis-free survival and relapse-free survival(secondary endpoints) in molecular subgroups, determined by the established MammaPrint, BluePrint, Targetprint and Theraprint profiles in addition to possible novel expression profiles.

DETAILED DESCRIPTION:
This will be a prospective observational, case-only study linking MammaPrint, BluePrint, TargetPrint, TheraPrint and possible additional profiles of interest to treatment response and Distant Metastases Free Survival (DMFS) and Relapse Free Survival (RFS). Only patients who receive neo-adjuvant therapy can participate.

For this project, approximately 50-70 institutions in the US will be invited to contribute clinical patient data from enrolled patients after a MammaPrint, TargetPrint, BluePrint and TheraPrint test has been successfully performed and the patient has started neo-adjuvant therapy.

Treatment is at the discretion of the physician, adhering to NCCN approved regimens or a recognized alternative.

The clinical data is to be entered online at 4 time points; amounting to four Case Report Forms (CRFs). Data will be collected on an ongoing basis, the first CRF must be completed within 6 weeks after the MammaPrint, BluePrint, TargetPrint, and TheraPrint result was provided. The second CRF should be completed 4 weeks after definitive surgery. CRF 3 and CRF4 will be completed 2-3 and 5 years after surgery.

It is expected that we will enroll around 1000 patients in 4 years.

OBJECTIVES

* Measure chemosensitivity (as defined by pCR) or endocrine sensitivity (as defined by decrease in longest tumor diameter or RCB1)in the molecular subgroups as determined by combining MammaPrint and BluePrint results.
* Correlate chemosensitivity (as defined by pCR) to TheraPrint Therapy Gene Assay results.
* Compare local IHC and FISH results (if available) with TargetPrint results. Compare the three BluePrint molecular subgroups with IHC-based subtype classification.
* Document impact of MammaPrint, TargetPrint and BluePrint result on treatment decision.
* Assess the 2-3 and 5 years DMFS and RFS for the different molecular subgroups.
* Measure chemosensitivity or endocrine sensitivity correlation with novel expression profiles.

ELIGIBILITY:
Inclusion Criteria:

* Women with histologically proven breast cancer, who have started or are scheduled to start neo-adjuvant chemotherapy therapy or neo-adjuvant hormone therapy, after successful MammaPrint assay
* Age 18-90
* Written informed consent

Exclusion Criteria:

* Patients who have had excisional biopsy or axillary dissection Patients with confirmed distant metastatic disease
* Tumor sample shipped to Agendia with ≤ 30% tumor cells or that fails QA or QC criteria
* Patients who have had any prior chemotherapy, radiotherapy, or endocrine therapy for the treatment of breast cancer
* Any serious uncontrolled intercurrent infections, or other serious uncontrolled concomitant disease

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with histologically proven breast cancer, who have started or are scheduled to start neo-adjuvant chemotherapy therapy or neo-adjuvant hormone therapy.
Sampling Method: Non-Probability Sample
Enrollment: 1142 (Actual)
Dates: Start 2011-07; Primary Completion 2015-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Chemosensitivity as defined by pCR | Up to 6 months
  For neo-adjuvant chemotherapy patients the primary endpoint is pathological complete response (pCR) which is defined as the absence of invasive carcinoma in both the breast and axilla at microscopic examination of the resection specimen, regardless of the presence of carcinoma in situ. The response rate and corresponding confidence intervals will be presented as a proportion of all patients enrolled. Comparison of response rates between different molecular subgroups will be conducted using Pearson Chi-square test.
Endocrine sensitivity as defined by partial response (decrease in longest tumor diameter or residual cancer burden category 1 (RCB1) | Up to 6 months
  The primary endpoint for patients with neo-adjuvant hormonal therapy is partial response which is defined as decrease in longest tumor diameter. The response rate and corresponding confidence intervals will be presented as a proportion of all patients enrolled. Comparison of response rates between different molecular subgroups will be conducted using Pearson Chi-square test.

SECONDARY OUTCOMES:
Correlate chemosensitivity (as defined by pCR) to TheraPrint Therapy Gene Assay results. | Up to 6 months.
  Correlation of chemosensitivity and endocrine sensitivity (as defined by pCR) to TheraPrint Therapy Gene Assay results will be determined using Pearson correlation and linear fit models.
Assess metastasis-free survival and relapse-free survival in molecular subgroups, determined by the established MammaPrint, BluePrint, profiles. | At -2-3 years and 5 years after definitive surgery.
  Kaplan-Meier curves for DMFS will be calculated for the following eight subgroups
  1. Luminal subtype
  2. ERBB2 subtype
  3. Basal subtype
  4. Luminal subtype and high risk MammaPrint
  5. Luminal subtype and low risk MammaPrint
  6. ERBB2 subtype and high risk MammaPrint
  7. ERBB2 subtype and low risk MammaPrint
Compare local IHC and FISH results (if available) with TargetPrint results. | Baseline; before start of neo-adjuvant therapy.
  Correlation of TargetPrint ER, PR, and HER2 microarray readout with IHC/FISH assessment will be determined using Pearson correlation and linear fit models. Agreement measurements between binary microarray and IHC classifications will be based on 2-way contingency table analysis and include overall concordance, positive agreement defined as the number of samples classified positive by both IHC and TargetPrint divided by the number of positive samples using IHC, negative agreement and Cohen's Kappa coefficient score.
Compare the three BluePrint molecular subgroups with IHC-based subtype classification. | Baseline; before start of neo-adjuvant therapy.
  Correlation of BluePrint molecular subgroup microarray readout with IHC-based subtype classification.
Document impact of MammaPrint, TargetPrint and BluePrint result on treatment decision. | Baseline; before start neo-adjuvant therapy.
  Review the impact of MammaPrint, TargetPrint, and BluePrint on physician treatment decisions.

CONTACTS AND LOCATIONS:
Overall Officials: Pat Whitworth, MD, Principal Investigator — Nashville Breast Center; Stephanie Akbari, MD, Principal Investigator — Reinsch Pierce Family Center for Breast Health; Mark Gittleman, MD, Principal Investigator — Breast Care Specialists; Peter Beitsch, MD, Principal Investigator — Dallas Surgical Group
Locations (75):
- United States (75):
  - Arizona Center for Cancer Care, Glendale, Arizona
  - 21 Century Oncology, Scottsdale, Arizona
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - Fresno Breast Surgery, Fresno, California
  - BreastLink, Long Beach, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - Community Hospital of Monterey Peninsula, Monterey, California
  - Alta Bates, Oakland, California
  - Comprehensive Cancer Center - Palm Springs, Palm Springs, California
  - Sutter Roseville Medical Center, Roseville, California
  - SHARP Memorial, San Diego, California
  - Redwood Regional, Santa Rosa, California
  - Wellness Oncology Hematology, West Hills, California
  - Exempla Health St Joseph, Denver, Colorado
  - Greenwich Hospital, Greenwich, Connecticut
  - Stamford Hospital, Stamford, Connecticut
  - Halifax Health Center for Oncology, Daytona Beach, Florida
  - Florida Hospital Memorial Medical Center, Daytona Beach, Florida
  - 21st Century Oncology, Fort Myers, Florida
  - St. Vincent Healthcare, Jacksonville, Florida
  - The Breast Institute at JFK Medical Center, Lake Worth, Florida
  - Baptist Health South Florida, Miami, Florida
  - Lakes Research, Miami Lakes, Florida
  - Dekalb Medical, Decatur, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Center for Breast Care, Savannah, Georgia
  - Advanced Breast Care Specialists, Bloomingdale, Illinois
  - University Surgical Consultants, Elk Grove Village, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Hematology/Oncology of The North Shore, Skokie, Illinois
  - Evansville Surgical Associates, Evansville, Indiana
  - Northern Indiana Cancer Research, South Bend, Indiana
  - Willis-Knighton Cancer Center, Shreveport, Louisiana
  - Signature Breast Care, Lanham, Maryland
  - McLaren Health Care, Burton, Michigan
  - Great Lakes Cancer Management Specialists, Grosse Pointe Woods, Michigan
  - Providence Cancer Institute, Southfield, Michigan
  - St Lukes Cancer Center, Kansas City, Missouri
  - Christian Hospital, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Compehensive Cancer Care of Nevada, Las Vegas, Nevada
  - Virtua Health, Willingboro, New Jersey
  - Ashikari Breast Center, Cortlandt Manor, New York
  - Hematology Oncology Associates of Central New York, East Syracuse, New York
  - Theresa & Eugene M. Lang Research Center, Flushing, New York
  - Akron General Hospital, Akron, Ohio
  - University of Toledo, Toledo, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Breast Care Specialists, Allentown, Pennsylvania
  - ACMH Cancer Center, Kittanning, Pennsylvania
  - St. Mary Medical Center, Langhorne, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - St. Clair Hospital, Pittsburgh, Pennsylvania
  - The Breast Place, Charleston, South Carolina
  - Cancer Specialists of Charleston, Charleston, South Carolina
  - Coastal Carolina Breast Center, Murrells Inlet, South Carolina
  - Nashville Breast Center, Nashville, Tennessee
  - Texas Tech University, Amarillo, Texas
  - Austin Cancer Center, Austin, Texas
  - Dallas Surgical Group, Dallas, Texas
  - Texas Health, Dallas, Texas
  - McAllen Oncology, Edinburg, Texas
  - East Houston General Surgery, Houston, Texas
  - Kathryn A. Wagner Private Practice, San Antonio, Texas
  - Radiation Oncology of San Antonio, San Antonio, Texas
  - Virginia Breast Care, Charlottesville, Virginia
  - Rockingham Memorial Hospital, Harrisonburg, Virginia
  - Lynchburg Hematology Oncology Clinic, Lynchburg, Virginia
  - Bon Secours Virginia Breast Center, Midlothian, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - Rockwood Clinic, Spokane, Washington
  - Bellin Hospital, Green Bay, Wisconsin
  - Columbia St. Marys Cancer Center, Milwaukee, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Wheaton Franciscan Healthcare, Wauwatosa, Wisconsin

REFERENCES:
- [Derived] Whitworth PW, Beitsch PD, Murray MK, Richards PD, Mislowsky A, Dul CL, Pellicane JV, Baron PL, Rahman RL, Lee LA, Dupree BB, Kelemen PR, Ashikari AY, Budway RJ, Lopez-Penalver C, Dooley W, Wang S, Dauer P, Menicucci AR, Yoder EB, Finn C, Blumencranz LE, Audeh W. Genomic Classification of HER2-Positive Patients With 80-Gene and 70-Gene Signatures Identifies Diversity in Clinical Outcomes With HER2-Targeted Neoadjuvant Therapy. JCO Precis Oncol. 2022 Sep;6:e2200197. doi: 10.1200/PO.22.00197. PMID 36108259
- [Derived] Whitworth PW, Beitsch PD, Pellicane JV, Baron PL, Lee LA, Dul CL, Murray MK, Gittleman MA, Budway RJ, Rahman RL, Kelemen PR, Dooley WC, Rock DT, Cowan KH, Lesnikoski BA, Barone JL, Ashikari AY, Dupree BB, Wang S, Menicucci AR, Yoder EB, Finn C, Corcoran K, Blumencranz LE, Audeh W; NBRST Investigators Group. Distinct Neoadjuvant Chemotherapy Response and 5-Year Outcome in Patients With Estrogen Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative Breast Tumors That Reclassify as Basal-Type by the 80-Gene Signature. JCO Precis Oncol. 2022 Apr;6(1):e2100463. doi: 10.1200/PO.21.00463. PMID 35476550